CLINICAL TRIAL: NCT04753736
Title: Intrauterine Administration and Immunophenotyping of Autologous Peripheral Blood Mononuclear Cells in Patients With Repeated Implantation Failures During Undergoing in Vitro Fertilization Treatment
Brief Title: Immunophenotypage of RIF and RM Patients and Intrauterine Administration of PBMC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of staff
Sponsor: Fertilys (Industry)
Collaborators: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Immunophenotypage RIF and RM
Record Dates: First submitted 2021-02-11; First posted 2021-02-15 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No recurrent implantation failure (No Intervention)
- Recurrent implantation failures (Experimental)
  Interventions: Procedure: Intrauterine administration of hCG-activated peripheral blood mononuclear cells
- Recurrent miscarriage (Experimental)
  Interventions: Procedure: Intrauterine administration of hCG-activated peripheral blood mononuclear cells

INTERVENTIONS:
Procedure: Intrauterine administration of hCG-activated peripheral blood mononuclear cells — Intrauterine administration of hCG-activated peripheral blood mononuclear cells
  Arms: Recurrent implantation failures; Recurrent miscarriage

SUMMARY:
The purpose of this study is to identify a systemic immunological profile specific to patients with recurrent implantation failures (RIF) or miscarriages (RM) through blood immunophenotyping on the day of ovulation. This study also aims to determine whether the intrauterine administration of 5 million peripheral blood monocluear cells increases implantation and pregnancy rates in patients with RIF and decreases the risk of miscarriages in patients with RM, compared to what has already been published in the scientific literature

ELIGIBILITY:
Inclusion Criteria:

* All women aged 18 and over undergoing an IVF cycle with her partner's sperm at the Fertilys fertility center, without a RIF status, agreeing to participate in the study and having signed the consent form to participate in the study.
* All women aged 18 and over undergoing an IVF cycle with her partner's sperm at the Fertilys fertility center, with a RIF or RM status, agreeing to participate in the study and having signed the consent form to participate in the study.

Exclusion Criteria:

* Women who need a gametes donor (eggs and / or sperm).
* Women undergoing an IVF cycle with frozen sperm.
* Women with autoimmune disease.
* Women with diabetes.
* Women with a history of chemotherapy treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-24 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Embryo implantation rate (biochemical pregnancy) | Two weeks following embryo transfer or 3 weeks following intrauterine insemination
Clinical pregnancy rate | Six to 8 weeks of gestation

SECONDARY OUTCOMES:
Peripheral blood mononuclear cells populations (PBMC) distribution at Day 0 | The day 0 of the patient's ovulation
Peripheral blood mononuclear cells populations distribution at Day 2 | After 48 hours of culture
Cytokines (LIF, IL-6, IL-10, TNFα, FGF-2, VEGF, IL-8) quantification by ELISA in PBMC culture medium at Day 2 | After 48 hours of culture

CONTACTS AND LOCATIONS:
Locations (1):
- Fertilys, Laval, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided